CLINICAL TRIAL: NCT02035085
Title: This is a First-in-man, Phase I Study Utilizing 19F Magnetic Resonance Imaging (MRI) to Track Autologous, Adipose Derived Stem Cells.
Brief Title: 19F Hot Spot MRI of Human Adipose-derived Stem Cells for Breast Reconstruction
Acronym: CS-1000
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drugs/devices discontinued
Sponsor: Johns Hopkins University (Other)
Collaborators: Cosmeticsurg.net (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00086592
Record Dates: First submitted 2013-12-19; First posted 2014-01-14 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: 19F MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CS-1000 (Experimental): Breast cancer patients with RIF will undergo liposuction, the autologous SVF cell fraction will be isolated and labeled with CS-1000 in the operating room without entering cell culture, which will then be returned to the patient at the site of breast grafting.
  Interventions: Drug: CS-1000 labeled SVF cells

INTERVENTIONS:
Drug: CS-1000 labeled SVF cells — Patients will undergo autologous transplantation of CS-1000 labelled SVF cells in a sterile environment.

SUMMARY:
Six female patients (>18 years of age, pre-menopausal) who have had loco-regional (lumpectomy and radiation) therapy for breast carcinoma and have been at least one-year disease free will undergo liposuction, the autologous SVF cell fraction will be isolated and labeled with CS-1000 in the operating room without entering cell culture, which will then be returned to the patient at the site of breast grafting. Patients will receive a pre-screening MRI . Patients will have an MRI scans over a period of 1 month at Johns Hopkins. Follow-up MRIs at 6,12, and 18 months will also be performed. Only at Johns Hopkins with fluorine being done as part of this investigational study. By performing fluorine MRI and quantification of 19F signal, we hypothesize that the engraftment of transplanted cells can be tracked in ways not possible before, using the total fluorine signal as surrogate marker for cell persistence and survival. We expect that a clinically successful outcome (maintenance of breast contour and volume) will be positively correlated with cell survival. The outcome of this study may pave the way for using 19F MRI cell tracking as a new tool for stem cell therapy in a variety of clinical applications.

ELIGIBILITY:
Inclusion Criteria:

1. Patient capable and willing to sign the Informed Consent (see attached document)
2. Patient must be willing to complete all visits in this study
3. Female, >18 years of age
4. Lumpectomy and radiation therapy for breast carcinoma
5. 18 month disease free survival
6. No evidence of metastatic disease
7. Patient is fit for surgery as determined by preoperative medical clearance workup performed by an independent primary care physician.
8. Negative pregnancy test.

Exclusion Criteria:

1. Evidence of metastatic disease
2. Less than 18 months disease-free interval
3. Unable to undergo MRI:

3a) Metallic implant 3b) Claustrophobic 4) High risk for surgical intervention because of comorbidities 5) Received treatment with an investigational drug within 30 days of screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
19F MRI signal over time | within 18 months
  The engraftment of transplanted cells will be tracked in ways not possible before, using the total fluorine signal as surrogate marker for cell persistence and survival.

SECONDARY OUTCOMES:
Maintenance of breast contour and volume | within 18 months
  CTCAE/CTEP scale examination criteria (retraction, atrophy, breast and arm edema, ulceration, telangiectasia, and induration/fibrosis will be used for assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff WM Bulte, PhD, Principal Investigator — Johns Hopkins University; Ricardo Rodriguez, MD, Study Director — Cosmeticsurg.net
Locations (1):
- CosmeticSurg, Lutherville-Timonium, Maryland, United States

REFERENCES:
- [Derived] Rose LC, Kadayakkara DK, Wang G, Bar-Shir A, Helfer BM, O'Hanlon CF, Kraitchman DL, Rodriguez RL, Bulte JW. Fluorine-19 Labeling of Stromal Vascular Fraction Cells for Clinical Imaging Applications. Stem Cells Transl Med. 2015 Dec;4(12):1472-81. doi: 10.5966/sctm.2015-0113. Epub 2015 Oct 28. PMID 26511652